CLINICAL TRIAL: NCT04493658
Title: Differential Diagnosis of Sjögren's Versus Non-Sjögren's Dry Eye
Status: Completed | Type: Observational
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Other Study IDs: IRB00247104
Record Dates: First submitted 2020-07-10; First posted 2020-07-30 (Actual); Last update posted 2023-01-05 (Actual); Status verified 2023-01

CONDITIONS: Keratoconjunctivitis Sicca; Dry Eye Syndromes; Ocular Surface Disease; Sjogren's Syndrome
Keywords: dry eye; keratoconjunctivitis sicca; ocular surface disease; sjogrens syndrome
MeSH Terms: conditions — Keratoconjunctivitis Sicca; Dry Eye Syndromes; Sjogren's Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Tear fluid samples and impression cytology
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Sjogrens syndrome dry eye: Patients with a previous diagnosis of dry eye made by an eye care specialist and a diagnosis of Sjogren's syndrome made according to the 2016 revised criteria
  Interventions: Diagnostic Test: Questionnaires; Diagnostic Test: Tear fluid sampling; Diagnostic Test: Impression Cytology
- Non-Sjogrens syndrome dry eye: Patients with a previous diagnosis of dry eye made by an eye care specialist and no diagnosis of Sjogren's syndrome based on 2016 revised criteria.
  Interventions: Diagnostic Test: Questionnaires; Diagnostic Test: Tear fluid sampling; Diagnostic Test: Impression Cytology
- Control: Normal individuals with no previous diagnosis of dry eye or Sjogren's syndrome
  Interventions: Diagnostic Test: Questionnaires; Diagnostic Test: Tear fluid sampling; Diagnostic Test: Impression Cytology

INTERVENTIONS:
Diagnostic Test: Questionnaires — Cognitive ability questionnaires, dry eye symptom questionnaires (Ocular Surface Disease Index, Impact of Dry Eye in Everyday Life, Visual Function Questionnaire-25, Eye Dryness Visual Analog Scale, Visual Fatigue Visual Analog Scale, Visual Tasking Questionnaire, Short Form Survey-36, Profile of Fatigue and Discomfort, European League Against Rheumatism Sjögren's Syndrome Patient Reported Index) will be completed by the subjects
Diagnostic Test: Tear fluid sampling — Using microcapillary tubes, 1 microliter of tear fluid will be collected in both eyes of each subject.
Diagnostic Test: Impression Cytology — Under topical anesthesia, impression cytology sampling will be performed in the temporal bulbar conjunctiva of both eyes of each subject.

SUMMARY:
To investigate and compare the burden of dry eye in Sjögren's syndrome dry eye vs non-Sjögren's syndrome dry eye, as well as investigate the diagnostic potential of tear film mucins and various inflammatory cytokines evaluated by tear fluid analysis and impression cytology.

DETAILED DESCRIPTION:
Dry eye is a prevalent ocular disorder worldwide and recognized as one of the most frequent reasons for seeking eye care. Whether locally or systemically initiated, inflammation plays a key role in the pathogenesis of dry eye. Approximately half of the patients with clinically significant dry eye have an underlying systemic inflammatory or autoimmune disease. One serious disease that causes significant dry eye is Sjögren's syndrome (SS). SS is an autoimmune disorder characterized by immune-mediated destruction of the salivary and lacrimal glands, with subsequent development of sicca symptoms. It is one of the most common autoimmune diseases in adults, affecting 1% to 4% of the general population. Approximately 10% of patients with clinically significant dry eye have underlying SS. Currently, the diagnosis of SS among dry eye patients is delayed by about a decade, largely due to lack of awareness and also diversity of patient symptoms and signs, adding to the complexity of diagnosis. Importantly, patients with SS are at risk for many ocular and systemic complications including central nervous system and visceral organ involvement as well as lymphoma. In fact, SS is the autoimmune disease most frequently associated with lymphoma. Therefore, identifying the subset of dry eye patients with SS is relevant.

Diagnosis of SS remains challenging mainly due to the lack of definitive diagnostic tests. The presence of aqueous-deficient dry eye is an integral part of diagnostic criteria for SS. Arguably, the hallmark of SS-related dry eye is conjunctival vital dye staining related to loss or alteration of the ocular surface mucins. A healthy conjunctiva is essential for ocular surface health as conjunctival goblet cells are responsible for secretion of the large gel-forming mucin MUC5AC which plays an important role in maintenance of the tear film on the ocular surface. Reduction of MUC5AC levels in tears of patients with SS has been demonstrated in a single previous study. The investigators also found lower levels of tear MUC5AC, and higher levels of IL-6 an IL-8 in patients with SS-dry eye in comparison to non-SS dry eye and controls. In addition, the investigators found the conjunctival lissamine green staining has a role in differentiating SS versus non-SS dry eye, independently of the dry eye severity.

In addition, increased levels of cytokines such as interleukin (IL)-13, IL-21, and interferon-gamma (IFN-γ) in tears and conjunctiva have previously been shown to correlate with goblet cell loss in SS as well as non-SS-dry eye patients. In murine studies, IFN-γ and tumor necrosis factor alpha (TNF-α) were reported to inhibit MUC5AC secretion in goblet cells stimulated with a cholinergic agonist. Such inhibition correlated with the expression of inflammatory cytokines in the conjunctiva of a mouse model of SS and significantly reduced tear MUC5AC levels. Nevertheless, targeting tear and ocular surface mucins and the relationships to various cytokines in dry eye as a diagnostic or therapeutic area has yet to be extensively studied.

Furthermore, it is well known that patients with SS-related dry eye have much more significant visual complaints than ocular discomfort symptoms arguably due to high corneal punctate erosion scores and diminished corneal subbasal nerve plexus when compared with non-SS dry eye patients. Although the exact mechanism of this is not known, cytokine levels in the tear film might possibly be a contributing factor. Indeed, the worsening of the corneal staining after prolonged gazing, could possibly be attributable to lack of tear film mucin as the investigators demonstrated the correlation between the conjunctival lissamine green staining (a surrogate for goblet cell density which secrete the mucin).

Lastly, although the advent of targeted biological treatments and other factors has led to renewed interest in Sjögren's among rheumatologists and immunologists, its ocular manifestations and burden remain underappreciated. As an example, the most widely used Sjögren's disease activity tool, the EULAR Sjögren's Syndrome Disease Activity Index (ESSDAI), does not include the extraglandular ocular manifestations of Sjögren's, such as corneal melt/perforation, uveitis, scleritis, retinal vasculitis, and optic neuritis. In addition, the EULAR Sjögren's Syndrome Patient Reported Index (ESSPRI) only includes one item that addresses the severity of dryness, but this refers to overall dryness and not specifically ocular dryness. Most importantly, these tools do not include any visual symptoms related to dry eye, such as blurred vision and visual or ocular fatigue. The investigators' most recent study points to a significant toll that the ocular manifestations of Sjögren's can have on patients emotionally, physically, and financially, in fact much more pronounced than other manifestation.

ELIGIBILITY:
Inclusion Criteria:

* Capacity to give informed consent
* Self-reported literacy
* Best corrected visual acuity at distance 20/40 in each eye
* Signed Institutional Review Board (IRB) approved consent agreeing to terms of the study

  * Additional inclusion criteria for the dry eye group (both SS- and non-SS) will include a previous diagnosis of dry eye made by an eye care specialist.
  * Differentiation of SS-related versus non-SS dry eye will be made according to the 2016 revised SS classification criteria.

The classification criteria are based on the weighted sum of the below 5 items:

• SS laboratory findings

* Anti-Sjogren's Antibody A (SSA) antibody positivity
* Focal lymphocytic sialadenitis with a focus score ≥ 1 foci/mm2

each scoring=3

• SS clinical findings

* Abnormal ocular staining score ≥ 5 (or van Bijsterveld score ≥ 4) in one eye
* Schirmer test ≤ 5 mm/5 min (without anesthesia) in one eye
* Unstimulated salivary flow rate ≤ 0.1 mL/min

each scoring=1

Individuals who have a total score ≥ 4 for the items above, meet the criteria for primary SS. In other words, for final classification, an individual should have at least one laboratory and one clinical finding.

Additional inclusion criteria for control subjects will include no previous history of dry eye diagnosis, and no known history of autoimmune disease, verified using a review of systems and past medical history form.

Exclusion Criteria:

* Age less than 18 years
* Known diagnoses of: Hepatitis C infection, HIV infection, Sarcoidosis, Amyloidosis, Graft Versus Host Disease (GVHD), Cicatrizing conjunctivitis (ie. from trachoma, Stevens-Johnsons Syndrome (SJS), pemphigoid, drug induced pseudo-pemphigoid, or chemical burns, other severe ocular surface diseases such as atopic keratoconjunctivitis
* Physical or mental issues, illiteracy, language problems which might possibly interfere with reading ability or other condition that would preclude successful participation in this study
* Contact lens wear within 10 days of enrollment
* Any intraocular surgery (including cataract surgery) within the last 3 months
* Any minor ocular surgery including tear duct cauterization or plugs, within the last 30 days
* Any history of corneal surgery or cosmetic lid surgery in the past 12 months
* Best corrected vision worse than 20/40
* Pregnant or nursing
* Artificial tear use within 24 hours of study visit
* History of taking or current use of topical prescription eye drops (including, cyclosporine and steroids as well as any glaucoma eye drops).

  * Patients who are willing to discontinue their treatment for at least a period of 30 days can be placed on a "wash-out period" as per the discretion of the investigator and patient safety, and be eligible at the end of this period, given all other criteria have been met. Otherwise, patients on these medications will be excluded.
  * Any person treated with glaucoma drops in the past (more than 30 days ago) or who had glaucoma surgery (more than 12 months ago) can be included.

    * Additional exclusion criteria for control subjects will include previous history of dry eye diagnosis, or history of any known autoimmune, inflammatory or rheumatologic disease including but not limited to Sjögren's syndrome, rheumatoid arthritis, Lupus, mixed connective tissue disease, scleroderma. Also the above exclusion criteria apply to control subjects.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adult individuals, both male and female, who have been diagnosed with dry eye, as well as adult normal controls will be included.
Sampling Method: Non-Probability Sample
Enrollment: 92 (Actual)
Dates: Start 2021-01-11 (Actual); Primary Completion 2022-10-03 (Actual); Study Completion 2022-10-03 (Actual)

PRIMARY OUTCOMES:
Mood Questionnaire | Once per patient on the day of enrollment.
  The "Mood Questionnaire" is a self-administered, 7-item questionnaire to measure the mood status. The score ranges from 7 to 28, higher score indicating better mood. The mean and median score in Sjogren's related dry eye group will be compared to non-Sjogren's and normal control group statistically.
Center for Epidemiologic Studies Depression Scale (CES-D) | Once per patient on the day of enrollment.
  The "Center for Epidemiologic Studies Depression Scale (CES-D)" is a self-administered, 20-item questionnaire to measure the mood and behavioral status. The score ranges between 0 to 60, higher scores indicate the presence of worse symptomology. The mean and median score in Sjogren's related dry eye group will be compared to non-Sjogren's and normal control group statistically.
Ocular Surface Disease Index (OSDI) | Once per patient on the day of enrollment.
  The "Ocular Surface Disease Index (OSDI)" is a self-administered, 12-item questionnaire to measure the dry eye status.). The score ranges from 0 to 100, higher scores indicate the presence of worse symptomology. The mean and median score in Sjogren's related dry eye group will be compared to non-Sjogren's and normal control group statistically.
Visual Functioning Questionnaire-25 (VFQ-25) | Once per patient on the day of enrollment.
  The "Visual Functioning Questionnaire-25 (VFQ-25)" is a self-administered, 25-item questionnaire to measure the vision related quality of life. The score ranges from 0 to 100, higher scores indicate better functioning. The mean and median score in Sjogren's related dry eye group will be compared to non-Sjogren's and normal control group statistically.
Impact of Dry Eye on Everyday Life (IDEEL) | Once per patient on the day of enrollment.
  The "Impact of Dry Eye on Everyday Life (IDEEL)" is a self-administered, 57-item questionnaire to measure the impact of dry eye and dry eye treatments on quality of life. Scores for each dimension ranges from 0 to 100. Higher scores indicate less impact on daily activities/work/emotions; greater bother due to symptoms; greater satisfaction with treatment effectiveness; and less treatment-related bother or inconvenience. The mean and median score in Sjogren's related dry eye group will be compared to non-Sjogren's and normal control group statistically.
Visual Tasking Questionnaire (VTQ) | Once per patient on the day of enrollment.
  The "Visual Tasking Questionnaire (VTQ)" is a self-administered, 14-item questionnaire to measure the visual functioning status. The composite score for a visual function is defined as the mean response for the items listed for that visual function. The mean and median score in Sjogren's related dry eye group will be compared to non-Sjogren's and normal control group statistically.
36 Item Short Form Survey (SF-36) | Once per patient on the day of enrollment.
  The "36 Item Short Form Survey (SF-36)" is a self-administered, 36-item questionnaire to measure the self-perceived health status. Scoring ranges from 0 to 100. The lower score indicates higher disability. The mean and median score in Sjogren's related dry eye group will be compared to non-Sjogren's and normal control group statistically.
Profile of Fatigue and Discomfort (PROFAD) | Once per patient on the day of enrollment.
  The "Profile of Fatigue and Discomfort (PROFAD)" is a self-administered, 19-item questionnaire to measure the fatigue status. Scoring ranges from 0 to 28, with higher scores indicating worse functioning. The mean and median score in Sjogren's related dry eye group will be compared to non-Sjogren's and normal control group statistically.
EULAR Sjogren's Syndrome Patient Reported Index (ESSPRI) | Once per patient on the day of enrollment.
  The "EULAR Sjogren's Syndrome Patient Reported Index (ESSPRI)" is a self-administered, 3-item questionnaire to measure the dryness, fatigue, and pain status. Scores range from 0 to 30, with higher scores indicating higher severity. The mean and median score in Sjogren's related dry eye group will be compared to non-Sjogren's and normal control group statistically.
Visual Fatigue Analogue Scale (VFAS) | Once per patient on the day of enrollment.
  The "Visual Fatigue Analogue Scale (VFAS)" is a self-administered, single scale indication, measuring visual fatigue. The score ranges from 0 to 100, with higher score indicating worse fatigue. The mean and median score in Sjogren's related dry eye group will be compared to non-Sjogren's and normal control group statistically.
Visual Dryness Analogue Scale (VDAS) | Once per patient on the day of enrollment.
  The "Visual Dryness Analogue Scale (VDAS)" is a self-administered, single scale indication, measuring eye dryness. The score ranges from 0 to 100, with higher score indicating worse dryness. The mean and median score in Sjogren's related dry eye group will be compared to non-Sjogren's and normal control group statistically.

SECONDARY OUTCOMES:
Impression Cytology of Ocular Surface | Once per patient on the day of enrollment.
  Impression cytology samples will be stained using Hematoxiline & Eosin. Samples will be examined using a light microscope. Mean and median goblet cell counts per high power field in Sjogren's related dry eye group will be compared to non-Sjogren's and normal control group statistically.
Inflammatory markers of tear film | Once per patient on the day of enrollment.
  Tear film MUC5AC levels will be assessed with enzyme-linked immunosorbent assay (ng/mL), and cytokines [CXCL9, CXCL11, CXCL13, IL-1, IL-2, IL-6, IL-8, IL-10, IL-12, IL-17, IFN-gamma, and TNF-alpha] (ng/mL) will be measured using a Luminex assay in a masked fashion. The mean and median level in Sjogren's related dry eye group will be compared to non-Sjogren's and normal control group statistically.

CONTACTS AND LOCATIONS:
Overall Officials: Esen Akpek, MD, Principal Investigator — Johns Hopkins Univeristy
Locations (1):
- Wilmer Eye Insitute, Johns Hopkins School of Medicine, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Akpek EK, Wu HY, Karakus S, Zhang Q, Masli S. Differential Diagnosis of Sjogren Versus Non-Sjogren Dry Eye Through Tear Film Biomarkers. Cornea. 2020 Aug;39(8):991-997. doi: 10.1097/ICO.0000000000002299. PMID 32195754
- [Background] Shiboski CH, Shiboski SC, Seror R, Criswell LA, Labetoulle M, Lietman TM, Rasmussen A, Scofield H, Vitali C, Bowman SJ, Mariette X; International Sjogren's Syndrome Criteria Working Group. 2016 American College of Rheumatology/European League Against Rheumatism Classification Criteria for Primary Sjogren's Syndrome: A Consensus and Data-Driven Methodology Involving Three International Patient Cohorts. Arthritis Rheumatol. 2017 Jan;69(1):35-45. doi: 10.1002/art.39859. Epub 2016 Oct 26. PMID 27785888